CLINICAL TRIAL: NCT03519048
Title: Randomized Multicentric Comparative Study Between a Conventional and an Intensive Follow up Strategy After Treatment of a Head and Neck Squamous Cell Carcinoma
Brief Title: Multicentric Comparative Study Between a Conventional and an Intensive Follow up Strategy After Treatment of a Head and Neck Squamous Cell Carcinoma
Acronym: SURVEILL'ORL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A01254-49; 2017/2553 (Other: CSET number)
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional follow-up (Active Comparator): clinical examination with nasofibroscopy every 1-3 months first year post-treatment, every 2-4 months second year, every 4-6 months third year (mean of around 13 visits) and every 6 months thereafter. Low Dose Chest CTscan every year in patients with tobacco consumption history of > 20 pack-year. Panendoscopy plus CT-scan are performed in case of clinical symptoms or abnormal clinical exam.
  Interventions: Procedure: Nasofibroscopy; Other: Low Dose Chest CTscan; Procedure: Biopsy
- Intensive follow-up strategy (Experimental): adding to the conventional follow-up strategy , an annual head&neck and thoracic injected CT-scan and Lugol upper gastrointestinal endoscopy (the first performed 12 months after inclusion), annual whole body PET-CT (the first at 6 months after inclusion). These 3 exams are performed every year during 3 years after inclusion (i.e. 3 CT-scan, 3 digestive endoscopies and 3 PET-CT per patient). Clinical follow up will be conducted as in the conventional follow up group and panendoscopy or bronchoscopy will be performed if needed. After 3 years, patients will be followed by conventional follow-up.
  Interventions: Other: injected CT-scan; Other: whole body PET-CT; Procedure: Lugol upper gastrointestinal endoscopy; Procedure: Biopsy

INTERVENTIONS:
Procedure: Nasofibroscopy — every 1-3 months first year post-treatment, every 2-4 months second year, every 4-6 months third year (mean of around 13 visits) and every 6 months thereafter
  Arms: Conventional follow-up
Other: Low Dose Chest CTscan — every year in patients with tobacco consumption history of > 20 pack-year
  Arms: Conventional follow-up
Other: injected CT-scan — the first performed 12 months after inclusion
  Arms: Intensive follow-up strategy
Other: whole body PET-CT — annual whole body PET-CT (the first at 6 months after inclusion)
  Arms: Intensive follow-up strategy
Procedure: Lugol upper gastrointestinal endoscopy — the first performed 12 months after inclusion
  Arms: Intensive follow-up strategy
Procedure: Biopsy — In both arm, patient will have a confirmation biopsy in case of suspicion of relapse or second primary.

SUMMARY:
Phase III randomized trial to compare the efficacy in terms of overall survival of two follow-up strategies (conventional versus intensive) among smokers and/or alcohol drinkers patients, older than 35 year, in complete remission 2-4 months after treatment of head and neck squamous cell carcinoma Patients will be randomized after the post-treatment check-up (clinical examination and reference imaging including PET-CT for patients ≥ N2) performed 2 to 4 months after the end of treatment. The randomization ratio is 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged superior to 35 years
* Current or previous smokers (smoked more than 10 packs year) or alcohol drinkers (current or previous, more than 140 g alcohol per week) or both
* Histologically proven invasive HNSCC stage 0 to IVa, excluding T4b and nasopharynx. Patients with in situ carcinoma are eligible.
* Treated with curative intent
* Free of cancer at the post-treatment clinical and radiological examination (negative PET-CT for N≥2) at least 2 months after the end of the last treatment and no later than 4 months after. If there is a strong doubt of lack of complete remission (for example if more exams or longer follow-up are needed to affirm or deny complete remission), the patient is not eligible for the trial.
* Remark: Patients with several head and neck squamous cell carcinoma (concomitant or successive), all treated with curative intent and all in complete remission, are eligible.
* Agree to have a long term follow-up
* Signed informed consent
* Patient affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Pregnant or breastfeeding women
* Severe psychiatric condition that may inhibit protocol participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Impossibility to perform the planned exams of the intensive strategy
* Nasopharyngeal carcinoma
* Other malignancies within 5 years prior to randomization that needs followup by PET-scan or chest CT or head and neck CT/MRI
* Any disease that needs follow-up by regular upper digestive endoscopy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephane TEMAM, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No